CLINICAL TRIAL: NCT03348748
Title: Three Pilot Studies of Stereotactic Body Radiation Therapy (SBRT) and Surgery in Non-small Cell Lung Cancer
Brief Title: Stereotactic Body Radiation Therapy Followed by Surgery in Treating Patients With Stage I-IIIA Non-small Cell Lung Cancer
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I 50717; NCI-2017-01950 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 50717 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2017-11-15; First posted 2017-11-21 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Stage I Non-Small Cell Lung Cancer AJCC v7; Stage IA Non-Small Cell Lung Carcinoma AJCC v7; Stage IB Non-Small Cell Lung Carcinoma AJCC v7; Stage II Non-Small Cell Lung Cancer AJCC v7; Stage IIA Non-Small Cell Lung Carcinoma AJCC v7; Stage IIB Non-Small Cell Lung Carcinoma AJCC v7; Stage IIIA Non-Small Cell Lung Cancer AJCC v7
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiosurgery; Thoracic Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Study 1 (highest-dose of SBRT, surgery) (Experimental): Patients with stage I or II NSCLC in the peripheral lung undergo highest-dose of Stereotactic Body Radiation Therapy over a single treatment fraction on day 1. Patients then undergo thoracic surgery on day 28.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Drug: Stereotactic Body Radiation Therapy; Procedure: Thoracic Surgical Procedure
- Study 2 (lowest-dose of SBRT, surgery) (Experimental): Patients with stage I or II NSCLC in the central lung undergo lowest-dose of Stereotactic Body Radiation Therapy over a single treatment fraction on day 1. Patients then undergo thoracic surgery on day 28.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Drug: Stereotactic Body Radiation Therapy; Procedure: Thoracic Surgical Procedure
- Study 3 (lowest- or higher-dose of SBRT, surgery) (Experimental): Patients with stage IIIA NSCLC in the any lung location undergo lowest- or higher-dose of Stereotactic Body Radiation Therapy over a single treatment fraction on day 1. Patients then undergo thoracic surgery on day 28.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Drug: Stereotactic Body Radiation Therapy; Procedure: Thoracic Surgical Procedure

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Drug: Stereotactic Body Radiation Therapy — Undergo lowest-dose of SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy
  Arms: Study 2 (lowest-dose of SBRT, surgery)
Drug: Stereotactic Body Radiation Therapy — Undergo lowest- or higher-dose of SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy
  Arms: Study 3 (lowest- or higher-dose of SBRT, surgery)
Drug: Stereotactic Body Radiation Therapy — Undergo highest-dose of SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy
  Arms: Study 1 (highest-dose of SBRT, surgery)
Procedure: Thoracic Surgical Procedure — Undergo thoracic surgery
  Other Names: Chest Surgery; Thoracic Surgery; Thoracic Surgical Procedures

SUMMARY:
This pilot clinical trial studies the effects of stereotactic body radiation therapy followed by surgery in treating patients with stage I-IIIA non-small cell lung cancer. Stereotactic body radiation therapy is a method of radiation that uses imaging to precisely locate a tumor and then deliver very high radiation doses to the tumor site in order to limit normal tissue toxicity or damage.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and feasibility of combining single fraction stereotactic body radiation therapy (SBRT) followed by surgery, in thoracic malignancies.

SECONDARY OBJECTIVES:

I. To estimate overall survival (OS) and progression-free survival (PFS) after single fraction SBRT followed by surgery, in thoracic malignancies.

II. To define any differences in quality of life/toxicity following SBRT based on tumor location/stage/tumor type.

TERTIARY OBJECTIVES:

I. To assess changes in T cell mediated immunity following SBRT in thoracic malignancies.

OUTLINE: Patients are assigned to 1 of 3 studies.

STUDY 1: Patients with stage I or II non-small cell lung cancer (NSCLC) in the peripheral lung undergo highest-dose of SBRT over a single treatment fraction on day 1. Patients then undergo thoracic surgery on day 28.

STUDY 2: Patients with stage I or II NSCLC in the central lung undergo lowest-dose of SBRT over a single treatment fraction on day 1. Patients then undergo thoracic surgery on day 28.

STUDY 3: Patients with stage IIIA NSCLC in the any lung location undergo lowest- or higher-dose of SBRT over a single treatment fraction on day 1. Patients then undergo thoracic surgery on day 28.

After completion of study treatment, patients are followed up at 6, 9, and 12 months, every 6 months for 2 years, and then annually for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Have an Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Have histologically proven diagnosis of: non-small cell lung cancer (NSCLC) (stage I, II, or IIIa)

  * Neoadjuvant or induction chemotherapy or biological (immune, vaccine, etc.)therapy for stage IIIa is allowed
  * Chemotherapy for another invasive malignancy is permitted if it has been treated definitively and the patient has remained disease free for >3 years
* Participant is able to undergo surgery (planned lobectomy or wedge resection)

  * Specifically, the participant has been or will have been cleared for surgery at the time of enrollment; the surgeon can accept the baseline tests done within 45 days prior to SBRT to clear the patient for surgery
* Participants of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) during treatment
* Participant or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Contraindication to SBRT (this includes the inability to cooperate with any aspect of SBRT: such as the inability to lie still and breathe reproducibly)
* Previous radiotherapy to the volume of lung or mediastinum currently involved by tumor
* Previous surgery for this lung or mediastinum tumor
* Plans for the patient to receive other concomitant antineoplastic therapy (including standard fractionated radiotherapy, chemotherapy, biological therapy, vaccine therapy, and surgery) while on this protocol(does not apply to neoadjuvant therapy as in inclusion criteria) except at disease progression
* Patients with active systemic, pulmonary, or pericardial infection
* Pregnant or nursing female participants
* Unwilling or unable to follow protocol requirements
* Any condition which in the investigator?s opinion deems the participant ineligible
* Received an investigational agent within 30 days prior to enrollment
* Stage IIIb

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2021-07-12 (Actual); Study Completion 2025-12-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-related grade 3-5 adverse events assessed using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v)4.0 | Up to 10 weeks post-surgery
  Comparison will be made with published historical and contemporaneous rates of toxicity with standard of care therapy for each of the study groups.

SECONDARY OUTCOMES:
Overall survival | Up to 5 years
  Will be measured and compared with published historical and contemporaneous rates of toxicity with standard of care therapy for each of the study groups.
Progression free survival | Up to 5 years
  Will be measured and compared with published historical and contemporaneous rates of toxicity with standard of care therapy for each of the study groups.

OTHER OUTCOMES:
Change in the mediators of tumor antigen presentation, co-stimulatory molecules, and immune effector cell populations assessed using multicolor flow cytometry, immunohistochemistry, and enzyme-linked immunosorbent assay (ELISA) | Baseline up to 10 weeks post-surgery
  Defined as CD4+ and CD8+ T-cells, T-regulatory cells (CD4+CD25+FoxP3+), natural killer cells, monocytes, macrophages, dendritic cells and myeloid derived suppressor cells. The study groups will be compared with age, sex, and stage matched controls. Immunohistochemistry results, flow cytometry results and ELISA results will be tabulated as percent change pre/post-radiation, and pre/post-thoracic surgery. The effects of these interventions will be assessed using permutation paired t-test, with multiplicity adjustments to maintain a 10% false discovery rate. Adjusted effect sizes will be obtained
Factors associated with T cell immunity in pathologic specimens | After surgery
  Comparison will be made to similar, blinded samples from patients who received surgery alone (by means of standard Lung DSRG approval).
Incidence of adverse events assessed using the NCI CTCAE v4.0 | Up to 10 weeks post-surgery
  Will be stratified by type of surgery (wedge resection, lobectomy, open versus thoracoscopic, and pneumonectomy).

CONTACTS AND LOCATIONS:
Overall Officials: Anurag Singh, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States